CLINICAL TRIAL: NCT03880916
Title: Effects of Duloxetine on Postoperative Wound Complication of Total Knee Arthroplasty(TKA) in Central Sensitization Patient
Brief Title: Effects of Duloxetine on Postoperative Wound Complication of Total Knee Arthroplasty (TKA) in Central Sensitization Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KC18MESI0455
Record Dates: First submitted 2019-03-06; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Duloxetine
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine group (Experimental): 1. Phase I (preemptive): 2weeks before operation (30mg for 2weeks)
  2. Phase II (maintenance): 6weeks after operation (30mg for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)
  Interventions: Drug: Duloxetine; Drug: Placebo
- Placebo group (Placebo Comparator): 1. Phase I (preemptive): 2weeks before operation (Placebo for 2weeks)
  2. Phase II (maintenance): 6weeks after operation (Placebo for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)
  Interventions: Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 1. Phase I (preemptive): 2weeks before operation (30mg for 2weeks)
  2. Phase II (maintenance): 6weeks after operation (30mg for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)
Drug: Placebo — Phase I (preemptive): 2weeks before operation (Placebo for 2weeks) Phase II (maintenance): 6weeks after operation (Placebo for 6 weeks) plus routine pain control (celecoxib, pregabalin, acetaminophen/tramadol, oxycodone)

SUMMARY:
Postoperative wound complications such as wound dehiscence, skin necrosis, persistent wound drainage, delayed healing, and superficial skin infection could have devastating consequences, leading to arthroplasty failure and patient morbidity requiring additional operations and prolonging hospitalization with substantial burden in cost of care. Recently, interest and research on central sensitization (CS) have been increasing. CS is closely correlated with excessive pain. It has two main characteristics: allodynia and hyperalgesia. CS is an abnormal and intense enhancement of pain mechanism by the central nervous system. One of the mechanisms by which this excessive pain occurs in CS is reduced activation of descending inhibitory pathway associated with deficiency in pathways primarily in response to serotonin and norepinephrine. Serotonin plays an important role in normal wound healing by affecting the formation of neovascularization, inflammatory reactions, fibroblasts and tissue proliferation essential for wound healing. Norepinephrine is also closely related to wound healing by controlling chemotaxis of macrophage essential for normal wound healing. CS is a risk factor for the development of postoperative wound complication after primary Total Knee Arthroplasty (TKA). Preclinical models of central sensitization suggest that duloxetine is effective in the treatment. Investigators will compare the wound complication following TKA of central sensitization patients in duloxetine group (n=40) with those in non-duloxetine group (n=40). Investigators will classify the central sensitization patients by central sensitization inventory and divide the central sensitization patients in to 2 groups (duloxetine and non-duloxetine group) randomly. Investigators checks the wound complication after primary TKA and visual assessment scale at preoperative, postoperative 2 days and 1, 2,6,12 weeks. All participants will receive postoperative pain control after TKA using the same pain control regimen and wound dressing regimen except duloxetine.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty
* having medicare insurance
* Central sensitization inventory (CSI)> 40 (Central sensitization patient )

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Allergy or intolerance to study medications
* Patients with an American society of anesthesiologist (ASA) classification of IV (angina, congestive heart failure, dementia, cerebrovascular accident)
* Chronic gabapentin or pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Alcohol, drug abuser
* Narcotics addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03-30 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
The rates of wound complication | Change from baseline wound complication at postoperative 2 days, 1 week, 2 weeks, 6 weeks, 12 weeks
  wound dehiscence, suture granuloma, prolonged wound ooze occurring after postoperative day 5, significant hematoma formation, or surgical site infection recorded. Post-operative additional interventions included delayed discharge from hospital due to wound problem, additional outpatient clinic visits to examine the surgical wound, local application of antibiotic ointment, superficial wound debridement or suturing in the office, hematoma aspiration, prescription of antibiotics, or reoperation.
Hormone level | Change from baseline hormone level at postoperative 2, 6, 12 weeks
  Cortisol, Serotonin, Norepinephrine related with Central Sensitization and wound healing

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) score | Change from baseline VAS score at postoperative 2 days, 1, 2, 6, 12 weeks
  Pain evaluation, It will be measured on a scale of 10 points. Minimum point is 0 and maximum point is 10. Higher values represent a worse outcome.
Range of motion of the knee joint | Change from baseline range of motion at postoperative 2 days, 1, 2, 6, 12 weeks
  Range of motion

IPD SHARING:
Plan to Share IPD: No